CLINICAL TRIAL: NCT07198789
Title: Randomized, Double-Blind, Placebo-Controlled Crossover Clinical Trial to Evaluate the Effect of a Functional Low-Glycemic Index Carbohydrates Versus Standard Wholegrain Carbohydrates on Glycolipid Metabolism and Vascular Stress Markers in Subjects With Suboptimal Triglyceridemia
Brief Title: Randomized, Double-blind Crossover Trial Comparing Low-GI Functional vs. Standard Wholegrain Carbohydrates on Glycolipid Metabolism and Vascular Stress Markers in Adults With Suboptimal Triglyceridemia
Acronym: GLOW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Arrigo F.G. Cicero, MD, PhD, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PNRR_ONFOODS_LowCharb
Record Dates: First submitted 2025-09-21; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Prevention; Diabetes Prevention; Inflammation; Nutrition
Keywords: Low glycemic index; Low-GI diet; Triglycerides-Glucose Index; Low-glycemic index carbohydrates; Wholegrain carbohydrates; Altograno®
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Altograno® Bakery Foods (Active Comparator): Altograno® Pasta, Pizza and Flatbrad
  Interventions: Other: Altograno® Bakery Foods
- Standard Whole-Grain Bakery Foods (Placebo Comparator): Industrial standard whole-grain Pasta, Pizza and Flatbrad, in substitution of the same amount of carbohydrates usually eaten in a stabilized diet
  Interventions: Other: Standard Whole-Grain Bakery Foods

INTERVENTIONS:
Other: Altograno® Bakery Foods — Altograno® Pasta, Pizza and Flatbrad, in substitution of the same amount of carbohydrates usually eaten in a stabilized diet
  Arms: Altograno® Bakery Foods
Other: Standard Whole-Grain Bakery Foods — Industrial standard whole-grain Pasta, Pizza and Flatbrad, in substitution of the same amount of carbohydrates usually eaten in a stabilized diet
  Arms: Standard Whole-Grain Bakery Foods

SUMMARY:
Low-glycemic index (GI) carbohydrates help prevent type 2 diabetes and cardiovascular disease by reducing postprandial glucose, insulin spikes, inflammation, and triglyceride synthesis. They improve weight, lipid profiles, and vascular health. Our study will compare functional low-GI vs. standard wholegrain carbs in a Mediterranean diet to assess their effect on the Triglycerides-Glucose Index, a marker of metabolic and cardiovascular risk, in subjects with suboptimal triglyceride levels.

DETAILED DESCRIPTION:
The consumption of carbohydrates with a low glycemic index (GI) has emerged as a cornerstone in the dietary prevention of type 2 diabetes mellitus (T2DM) and cardiovascular disease (CVD). The glycemic index classifies carbohydrate-containing foods based on their impact on postprandial blood glucose: low-GI foods have a GI ≤ 55, medium-GI between 56 and 69, and high-GI ≥ 70. Low-GI foods cause slower and smaller rises in blood glucose and insulin, which can reduce glycemic variability and postprandial hyperglycemia.

Postprandial hyperglycemia is known to trigger oxidative stress and endothelial dysfunction, mechanisms closely involved in the pathogenesis of atherosclerosis and diabetic vascular complications. Clinical trials show that replacing high-GI carbohydrates with low-GI options improves fasting blood glucose by an average of 0.4 mmol/L and HbA1c by 0.3% in individuals with impaired glucose tolerance. These modest changes translate into meaningful reductions in the long-term risk of diabetes.

A pooled analysis of 24 prospective cohort studies found that a high-GI diet was associated with a 27% greater risk of developing T2DM. Moreover, each 5-unit increment in dietary GI increases the risk of coronary heart disease (CHD) by 13%. The metabolic advantage of low-GI carbohydrates lies in their ability to limit insulin spikes, reduce inflammatory cytokine release, and lower triglyceride synthesis.

In overweight individuals, low-GI diets are associated with greater weight loss and fat mass reduction than high-GI diets, even when total calories are similar. One study found that participants on a low-GI diet lost 1.5 kg more fat mass over 12 weeks compared to those on a high-GI diet, despite identical energy intake.

Low-GI foods also improve lipid profiles. A systematic review and meta-analysis reported a mean reduction of 0.13 mmol/L in LDL cholesterol and a 0.05 mmol/L increase in HDL cholesterol among participants consuming low-GI diets. These effects are particularly relevant in patients with metabolic syndrome or insulin resistance.

In children and adolescents, low-GI intake improves insulin sensitivity and reduces early markers of vascular damage. A randomized controlled trial demonstrated that adolescents on a low-GI diet exhibited lower carotid intima-media thickness (IMT), a surrogate marker of atherosclerosis progression, after six months.

Furthermore, a Mediterranean dietary pattern, which is naturally low in GI due to its emphasis on legumes, whole grains, and vegetables, has been linked to a 30% reduction in major cardiovascular events in high-risk populations. The PREDIMED trial showed that such a diet significantly reduced the incidence of myocardial infarction and stroke over five years.

Inflammation plays a central role in both T2DM and CVD, and low-GI diets help reduce C-reactive protein (CRP) levels by 0.5-1.0 mg/L on average. This anti-inflammatory effect may be one of the mechanisms through which low-GI diets offer cardiovascular protection.

Even among elderly individuals, adherence to low-GI diets has been associated with better cognitive function and glycemic control. A cross-sectional analysis showed that older adults in the highest tertile of dietary GI had significantly lower memory scores than those in the lowest tertile.

The combined effects of low-GI diets-improving glucose control, reducing inflammation, enhancing lipid profiles, and promoting satiety-make them an essential component of preventive nutrition strategies for chronic disease.

Public health guidelines increasingly recommend the substitution of refined carbohydrates with low-GI alternatives to curb the global diabetes epidemic. However, no direct comparison has been made so far between functional low-glycemic index carbohydrates and standard wholegrain carbohydrates in the context of a Mediterranean diet.

In this context, the primary purpose of our research will be to evaluate if functional low-glycemic index carbohydrates are able to reduce the Triglycerides-Glucose Index plasma levels versus standard wholegrain carbohydrates in healthy subjects with suboptimal triglycerides levels. The Triglycerides-Glucose Index is a cheap, validated, emerging risk factors for both metabolic and cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* TG>150 mg/dL
* Subjects who have the capability to communicate and to comply with the study's requirements.
* Subjects agree to participate in the study and having dated and signed the informed consent form.

Exclusion Criteria:

* Gluten hypersensitivity/Coeliac disease diagnosis
* BMI>30 kg/m2
* Any preventive treatments (i.e. lipid-lowering drugs, antihypertensives) not stabilized in type and dose for at least 3 months
* Any medical or surgical condition that would limit the patient adhesion to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Impact of Low-GI Functional Carbohydrates on TyG Index | 28 days
  To test whether functional low-glycemic index carbohydrates is able to reduce the Triglycerides-Glucose Index plasma levels versus standard wholegrain carbohydrates in healthy subjects

SECONDARY OUTCOMES:
Impact of Low-GI Functional Carbohydrates on Triglycerides | 28 days
  To test whether functional low-glycemic index carbohydrates is able to reduce the triglycerides plasma levels versus standard wholegrain carbohydrates in healthy subjects with suboptimal triglycerides levels
Impact of Low-GI Functional Carbohydrates on Fasting Glucose | 28 days
  To test whether functional low-glycemic index carbohydrates is able to reduce the fasting glucose plasma levels versus standard wholegrain carbohydrates in healthy subjects with suboptimal triglycerides levels
Impact of Low-GI Functional Carbohydrates on Non-HDL Cholesterol | 28 days
  To test whether functional low-glycemic index carbohydrates is able to reduce the Non-HDL cholesterol plasma levels versus standard wholegrain carbohydrates in healthy subjects with suboptimal triglycerides levels.
Impact of Low-GI Functional Carbohydrates on Apolipoprotein B | 28 days
  To test whether functional low-glycemic index carbohydrates is able to reduce the apolipoprotein B plasma levels versus standard wholegrain carbohydrates in healthy subjects with suboptimal triglycerides levels
Impact of Low-GI Functional Carbohydrates on hsCRP | 28 days
  To test whether functional low-glycemic index carbohydrates is able to reduce the hsCRP plasma levels versus standard wholegrain carbohydrates in healthy subjects with suboptimal triglycerides levels.
Impact of Low-GI Functional Carbohydrates on Endothelial Function | 28 days
  To test whether functional low-glycemic index carbohydrates is able to improve the endothelial function standard wholegrain carbohydrates in healthy subjects with suboptimal triglycerides levels.